CLINICAL TRIAL: NCT02577185
Title: An Exploratory Psoriasis Plaque Test Trial Investigating the Neurogenic Component in Psoriasis Vulgaris by Use of Botulinum Toxin A as Tool Compound
Brief Title: An Exploratory Trial Investigating the Neurogenic Component in Psoriasis Vulgaris by Use of Botulinum Toxin A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EXP-1187
Record Dates: First submitted 2015-10-09; First posted 2015-10-16 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin type A (Experimental): Experimental drug
  Interventions: Drug: Botulinum Toxin Type A
- sodium chloride 9 mg/ml (Placebo Comparator): Vehicle drug
  Interventions: Drug: Sodium chloride 9 mg/ml

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Arms: botulinum toxin type A
Drug: Sodium chloride 9 mg/ml
  Arms: sodium chloride 9 mg/ml

SUMMARY:
The purpose of this study is to evaluate the anti-psoriatic effect of injected Botulinum toxin type A compared to that of injected vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* A diagnosis of psoriasis vulgaris with lesions located on arms and/or legs and/or trunk
* Chronic stable psoriasis vulgaris diagnosed more than 6 months prior to screening.
* Women must use a reliable contraceptive during the trial.

Exclusion Criteria:

* Pregnant or breast feeding women, or women planning to become pregnant.
* Skin infection at injection sites
* Use of biological therapies or small molecules (marketed or not marketed) with a possible effect on psoriasis vulgaris
* Use of systemic treatments with a potential effect on psoriasis vulgaris
* Exposure to phototherapy within 4 weeks for PUVA and 2 weeks for UVB prior to Randomisation
* Use of potent or very potent (WHO group III-IV) corticosteroids for topical treatment of psoriasis within a 4 week period prior to randomisation
* Use of muscle relaxants
* History of dysphagia or aspiration
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Absolute change in Total Clinical Score (TCS) of clinical signs at 8 weeks after injection compared to baseline | 8 weeks

SECONDARY OUTCOMES:
Absolute change in clinical score erythema at week 1 compared to baseline | 1 week
Absolute change in clinical score erythema at week 3 compared to baseline | 3 weeks
Absolute change in clinical score erythema at week 4 compared to baseline | 4 weeks
Absolute change in clinical score erythema at week 8 compared to baseline | 8 weeks
Absolute change in clinical score scaling at week 1 compared to baseline | 1 week
Absolute change in clinical score scaling at week 3 compared to baseline | 3 weeks
Absolute change in clinical score scaling at week 4 compared to baseline | 4 weeks
Absolute change in clinical score scaling at week 8 compared to baseline | 8 weeks
Absolute change in clinical score infiltration at week 1 compared to baseline | 1 week
Absolute change in clinical score infiltration at week 3 compared to baseline | 3 weeks
Absolute change in clinical score infiltration at week 4 compared to baseline | 4 weeks
Absolute change in clinical score infiltration at week 8 compared to baseline | 8 weeks
Absolute change in TCS at week 1 compared to baseline | 1 week
Absolute change in TCS at week 3 compared to baseline | 3 weeks
Absolute change in TCS at week 4 compared to baseline | 4 weeks
Incidence of treatment emergent adverse events | 10 weeks
Incidende of adverse events on the treated test sites | 10 weeks
Incidence of adverse events leading to withdrawal from trial | 8 weeks
Change in blood pressure from baseline to week 8 | 8 weeks
Change in heart rate from baseline to week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Iversen, MD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Hud- og Kønssygdomme, Aarhus Universitetshospital, Aarhus
  - Hud- og allergiafdeling, Gentofte Hospital, Gentofte Municipality

IPD SHARING:
Plan to Share IPD: No